CLINICAL TRIAL: NCT05254002
Title: A Parallel-group Treatment, Phase 2, Double-blind, Three-arm Study to Assess Efficacy and Safety of Finerenone Plus Empagliflozin Compared With Either Finerenone or Empagliflozin Alone in Participants With Chronic Kidney Disease and Type 2 Diabetes.
Brief Title: A Study to Learn How Well the Treatment Combination of Finerenone and Empagliflozin Works and How Safe it is Compared to Each Treatment Alone in Adult Participants With Long-term Kidney Disease (Chronic Kidney Disease) and Type 2 Diabetes
Acronym: CONFIDENCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21839; 2023-506981-30-00 (Registry Identifier: CTIS); 2021-003037-11 (EudraCT Number)
Record Dates: First submitted 2022-02-04; First posted 2022-02-24 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes Mellitus; Chronic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — finerenone; empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Finerenone and Empagliflozin (Experimental): Participants will take Finerenone (10 or 20 mg once daily [OD]) and Empagliflozin (10 mg OD) for up to 180 days.
  Interventions: Drug: Finerenone (BAY94-8862 ) 10 mg; Drug: Empagliflozin; Drug: Finerenone (BAY94-8862 ) 20 mg
- Finerenone and Empagliflozin placebo (Experimental): Participants will take Finerenone (10 or 20 mg OD) and matching placebo to Empagliflozin (OD) for up to 180 days.
  Interventions: Drug: Finerenone (BAY94-8862 ) 10 mg; Drug: Empagliflozin Placebo; Drug: Finerenone (BAY94-8862 ) 20 mg
- Empagliflozin and Finerenone placebo (Experimental): Participants will take Empagliflozin (10 mg OD) and matching placebo to Finerenone (OD). for up to 180 days.
  Interventions: Drug: Empagliflozin; Drug: Finerenone Placebo

INTERVENTIONS:
Drug: Finerenone (BAY94-8862 ) 10 mg — oral administration, once daily if screening eGFR (Estimated glomerular filtration rate) results are: <60 mL/min/1.73 m2
  Arms: Finerenone and Empagliflozin; Finerenone and Empagliflozin placebo
Drug: Empagliflozin — oral administration, once daily
  Arms: Empagliflozin and Finerenone placebo; Finerenone and Empagliflozin
Drug: Empagliflozin Placebo — Matching placebo to empagliflozin oral administration, once daily
  Arms: Finerenone and Empagliflozin placebo
Drug: Finerenone (BAY94-8862 ) 20 mg — oral administration, once daily if screening eGFR (Estimated glomerular filtration rate) results are: ≥60 mL/min/1.73 m2
  Arms: Finerenone and Empagliflozin; Finerenone and Empagliflozin placebo
Drug: Finerenone Placebo — Matching Placebo to Finerenone oral administration once daily
  Arms: Empagliflozin and Finerenone placebo

SUMMARY:
Finerenone works by blocking a group of proteins, called mineralocorticoid receptor. An increased stimulation of mineralocorticoid receptor is known to trigger injury and inflammation in the kidney and is therefore thought to play a role in CKD.

Empagliflozin lowers blood sugar levels by increasing the excretion of glucose from the blood into the urine.

In this study, the researchers want to learn how well the combination of finerenone and empagliflozin helps to slow down the worsening of the participants' kidney function compared to either treatment alone. For this, the level of protein in the urine will be measured. The investigators also want to know how safe the combination is compared to either treatment alone.

Depending on the treatment group, the participants will either take the combination of finerenone and empagliflozin, or finerenone together with a placebo, or empagliflozin together with a placebo, once a day as tablets by mouth. A placebo looks like a treatment but does not have any medicine in it. Importantly, the participants will also continue to take their other current medicine for CKD and T2D.

The participants will be in the study for up to 7.5 months and will take the study treatments for 6 months. During the study, participants will visit the study site 7 times.

The study team will:

* collect blood and urine samples
* check the participants' vital signs
* do a physical examination including height and weight
* check the participants' heart health by using an electrocardiogram (ECG)
* monitor the participants' blood pressure
* ask the participants questions about how they are feeling and what adverse events they may be having An adverse event is any problem that happens during the trial. Doctors keep track of all events that happen in trials, even if they do not think the events might be related to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Participant with a clinical diagnosis of chronic kidney disease (CKD) and the following:

  * In Part A: eGFR 40-90 ml/min/1.73m^2 (with no more than 20% having an eGFR >75 ml/min/1.73m^2) using Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) formula at screening visit and at least one historical value of eGFR <60 mL/min/1.73 m^2 within 3 months or have a registered diagnosis of CKD.
  * In Part B: eGFR 30-90 ml/min/1.73m^2 (with no more than 20% having an eGFR >75 ml/min/1.73m^2) using CKD-EPI formula at screening visit and at least one historical value of eGFR <60 mL/min/1.73 m^2 within 3 months or have a registered diagnostic of CKD.
  * 100 ≤UACR <5000 mg/g at screening visit (mean value from 3 morning void samples) and documentation of albuminuria/proteinuria (quantitative or semi-quantitative measurement) in the participant's medical records at least 3 months prior to screening
* Participant with type 2 diabetes (T2D) as defined by the American Diabetes Association (ADA 2021), with glycated hemoglobin (HbA1c) at screening <11%.
* Participant treated with the clinically maximum tolerated dose, as per investigator judgment, of angiotensin-converting enzyme inhibitor (ACEi) or angiotensin receptor blocker (ARB), but not both, for more than 1 month at screening visit.

Exclusion Criteria:

* Participants with type 1 diabetes (T1D).
* Participant with hepatic insufficiency classified as Child-Pugh C.
* Participant with blood pressure at Day 1 visit (Visit 2) higher than 160 systolic blood pressure (SBP) or 100 diastolic blood pressure (DBP) or SBP lower than 90 mmHg.
* Participant currently treated with a sodium/glucose cotransporter-2 inhibitor (SGLT2i) or SGLT-1/2i or who received a SGLT2i or SGLT-1/2i which cannot be discontinued at least 8 weeks prior to the screening visit and during study intervention treatment.
* Participant treated with another mineralocorticoid receptor antagonist (MRA) (e.g., eplerenone, esaxerenone, spironolactone, canrenone), a renin inhibitor, potassium supplements, a potassium sparing diuretic (e.g., amiloride, triamterene), a potassium binder agent, or angiotensin receptor-neprilysin inhibitor (ARNI) which cannot be discontinued at least 8 weeks prior to the screening visit and during study intervention treatment.
* Participants currently treated or who were treated with Finerenone (Kerendia©) within 8 weeks prior to the screening visit.
* Participant with serum/plasma potassium (K+) above 4.8 mmol/L at screening visit (central laboratory value).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1664 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Relative change from baseline in UACR at 180 days in combination therapy group versus empagliflozin alone | Up to 180 days
  Urinary albumin to-creatinine ratio (UACR)
Relative change from baseline in UACR at 180 days in combination therapy group versus finerenone alone | Up to 180 days
Mean ratio of change from baseline to Day 180 in UACR for the combination therapy group, to empagliflozin alone | Upto 180 days
Mean ratio of change from baseline to Day 180 in UACR for the combination therapy group, to finerenone alone | Up to 180 days

SECONDARY OUTCOMES:
Relative change in UACR between end of treatment visit (Day 180) and 30 days after end of treatment visit (Day 210) | Up to 210 days
Relative change in UACR between 30 days after end of treatment visit (Day 210) and baseline (Day 1) | Up to 210 days
Relative change in UACR category (>30%, >40%, >50%) at 180 days | Up to 180 days
Ratio of change from baseline in eGFR at 30 days | Up to 30 days
  estimated glomerular filtration rate (eGRF)
eGFR decline greater than 30% at 30 days from baseline | Up to 30 days
Ratio of change in eGFR at 180 days and 210 days from Day 30 | Up to 210 days
Proportion of participants with of acute kidney injury (AKI) events | Up to 180 days
  AKI is defined as any of the following:
  * An increase in serum creatinine by greater than or equal to 0.3 mg/dL within 48 hours; or
  * An increase in serum creatinine by greater than or equal to 1.5 times baseline, which is known or presumed to have occurred within the prior 7 days; or
  * A urine volume less than 0.5 ml/kg/h for 6 hours
Total number of AKI events | Up to 180 days
Proportion of participants with hyperkalemia events (moderate hyperkalemia [5.5 <K+ ≤6.0 mmol/L], severe hyperkalemia [K+ >6.0 mmol/L]) | Up to 180 days
  serum/plasma potassium (k+)
Total number of hyperkalemia events (moderate hyperkalemia [5.5 <K+ ≤6.0 mmol/L], severe hyperkalemia [K+ >6.0 mmol/L]) | Up to 180 days
Change from baseline in K+ | Up to 180 days
Proportion of participants with severe hypoglycemia events | Up to 180 days
  Severe hypoglycemia is defined as glucose level of <3.0 mmol/L (<54 mg/dL).
Total number of events of severe hypoglycemia events | Up to 180 days
Proportion of participants with symptomatic hypotension events | Up to 180 days
Total number of symptomatic hypotension events | Up to 180 days
Proportion of participants with genital mycotic events | Up to 180 days
Total number of genital mycotic events | Up to 180 days
Proportion of participants with ketoacidosis events | Up to 180 days
Total number of ketoacidosis events | Up to 180 days
Proportion of participants with necrotizing fasciitis of the perineum events | Up to 180 days
Total number of necrotizing fasciitis of the perineum events | Up to 180 days
Proportion of participants with urosepsis and pyelonephritis events | Up to 180 days
Total number of urosepsis and pyelonephritis events | Up to 180 days

CONTACTS AND LOCATIONS:
Locations (185):
- United States (49):
  - Southwest Kidney Institute, PLC, Surprise, Arizona
  - Academic Medical Research Institute, Los Angeles, California
  - Northridge Hospital, Northridge, California
  - Olive View - UCLA Medical Center, Sylmar, California
  - Touro University California, Vallejo, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Florida Kidney Physicians - Delray Beach Nephrology, Delray Beach, Florida
  - West Orange Endocrinology & Clinical Research, Ocoee, Florida
  - Innovative Research Institute, Port Charlotte, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Grady Memorial Hospital - Endocrinology, Atlanta, Georgia
  - Southeast Kidney Associates, East Point, Georgia
  - Velocity Clinical Research - Savannah, Savannah, Georgia
  - Versailles Family Medicine, Versailles, Kentucky
  - Nola Care Clinical Research, Metairie, Louisiana
  - Omega Clinical Research Center, Metairie, Louisiana
  - South Shore Nephrology, Plymouth, Massachusetts
  - Lake Michigan Nephrology, Saint Joseph, Michigan
  - Clinical Research Consultants, Kansas City, Missouri
  - Kansas City VA Medical Center - Endocrinology, Kansas City, Missouri
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - St. Louis Heart & Vascular, PC, St Louis, Missouri
  - Somnos Clinical Research, Lincoln, Nebraska
  - Meridian Clinical Research- Norfolk, Norfolk, Nebraska
  - Healor Primary Care / CCT Research, Las Vegas, Nevada
  - Santa Rosa Medical Centers of Nevada / CCT Research, Las Vegas, Nevada
  - Circuit Clinical/Crystal Run, Middletown, New York
  - Randolph Medical Associates, Asheboro, North Carolina
  - University of North Carolina Kidney Center, Chapel Hill, North Carolina
  - Eastern Nephrology Associates - Greenville West, Greenville, North Carolina
  - Blue Sky, MD/ Lamond Family Medicine, Hendersonville, North Carolina
  - Eastern Nephrology Associates - Kinston, Kinston, North Carolina
  - Velocity Clinical Research, Cincinnati, Cincinnati, Ohio
  - Oakland Medical Center, Dakota Dunes, South Dakota
  - Dunes Clinical Research LLC, Dakota Dunes, South Dakota
  - DarSalud Care / LifeDOC Research, Memphis, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Office of Osvaldo A. Brusco, MD, Corpus Christi, Texas
  - Thyroid, Endocrinology, and Diabetes (TED) PA, Dallas, Texas
  - DaVita Clinical Research- El Paso, El Paso, Texas
  - Global Kidney Center, Houston, Texas
  - Victorium Clinical Research, Houston, Texas
  - North Texas Kidney Disease Associates, PLLC, Lewisville, Texas
  - Biopharma Informatic - McAllen, TX, McAllen, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - Olympus Family Medicine, Salt Lake City, Utah
  - Salem VA Medical Center - Endocrinology, Salem, Virginia
  - MultiCare Rockwood Clinic Diabetes & Endocrinology Center, Spokane, Washington
- Belgium (8):
  - CHU de Charleroi Hôpital civil, Lodelinsart, Hainaut
  - Onze-Lieve-Vrouwziekenhuis (OLVZ) - Campus Aalst, Aalst, Oost-vlaanderen
  - AZ St-Lucas Campus St-Lucas, Ghent
  - UZ Gent, Ghent
  - Regionaal ZH Jan Yperman Campus Mariaziekenhuis, Ieper
  - AZ Groeninge Campus Kennedylaan, Kortrijk
  - UZ Leuven Gasthuisberg, Leuven
  - AZ Delta, Roeselare
- Canada (9):
  - LMC Manna Research - Calgary, Calgary, Alberta
  - Hamilton Medical Research Group, Hamilton, Ontario
  - William Osler Health centre, Sakuara Medical, Mississauga, Ontario
  - Bluewater Clinical Research Group, Sarnia, Ontario
  - Sameh Fikry Professional Corporation, Waterloo, Ontario
  - Clinical Research Solutions, Inc., Waterloo, Ontario
  - Recherche GCP Research, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - LMC Clinical Research Inc. Montreal, Saint-Laurent, Quebec
- Denmark (4):
  - Bispebjerg Hospital - Hjerteafdeling, Copenhagen
  - Hospital of South West Jutland | Department of Endocrinology Research, Esbjerg
  - Steno Diabetes Center Copenhagen | Herlev - Clinical and Translational Research Department, Herlev
  - Region Midtjylland | Regionshospitalet Godstrup - Nephrology Department, Herning
- France (6):
  - Hôpital François Mitterrand - Dijon, Dijon
  - Center Hospitalier Michallon - Grenoble, Grenoble
  - Hôpital Edouard Herriot - Lyon Cedex, Lyon
  - Many Locations, Multiple Locations
  - Hopital Carémeau - Nîmes, Nîmes
  - Hôpital Saint Joseph, Paris
- Germany (8):
  - St. Josefskrankenhaus, Heidelberg, Baden-Wurttemberg
  - ClinPhenomics GmbH&Co. KG, Frankfurt am Main, Hesse
  - Diabetologische Schwerpunkt Praxis Dortmund, Dortmund, North Rhine-Westphalia
  - Zentrum für Diabetologie und Ernährungsmedizin, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Cardiologicum Pirna / Dresden-Seidnitz, Pirna, Saxony
  - Friedrich-Schiller-Uni. Jena, Jena, Thuringia
  - Charité Campus Benjamin Franklin (CBF), Berlin
  - Diabetes Zentrum Wandsbek, Hamburg
- India (26):
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - Mavani Dialysis & Kidney Center, Ahmedabad, Gujarat
  - K.L.E.S. Dr. Prabhakar Kore Hospital & Medical Research Centre, Belagavi, Karnataka
  - Manipal Hospital, Mysore, Karnataka
  - Asian Kidney Hospital and Medical Centre, Nagapur, Maharashtra
  - All India Institute of Medical Sciences, Bhubaneswar, National Capital Territory of Delhi
  - Indraprastha Apollo Hospital, New Delhi, National Capital Territory of Delhi
  - Eternal Heart Care Centre (EHCC) and Research Institute, Jaipur, Rajasthan
  - Osmania General Hospital, Telangana, Telangana
  - G.S.V.M. Medical College, Kanpur, Uttar Pradesh
  - Institute of Post-Graduate Medical Education and Research, Kolkata, West Bengal
  - Dr. Bantwal's Clinic, Bengaluru
  - Bangalore Medical College & Research Institute, Bengaluru
  - Government Kilpauk Medical College Hospital, Chennai
  - Sriram Chandra Bhanj Medical College & Hospital, Cuttack
  - Nizam's Institute of Medical Sciences (NIMS), Hyderabad
  - Sawami Man Singh (SMS) Medical College & Attached Hospitals, Jaipur
  - Government Medical College, Kozhikode
  - Vinaya Hospital and Research Centre (A Unit of KIMS), Mangalore
  - Seth Gordhandas Sunderdas Medical College (GSMC) - King Edward Memorial (KEM) Hospital, Mumbai
  - Government Medical College and Hospital (GMCH) Nagpur, Nagpur
  - Max Super Speciality Hospital (MSSH) - Saket, New Delhi
  - Grant Medical Foundation - Ruby Hall Clinic (RHC), Pune
  - Lifepoint Multispecialty Hospital, Pune
  - Krishna Institute Of Medical Science, Secunderabad
  - Vedanta Kidney Care, Vadodara
- Israel (8):
  - HaEmek Medical Center | Internal Medicine C Department - Research Unit, Afula
  - Barzilai Medical Center | Department of Nephrology and Hypertension, Ashkelon
  - Clalit Health | Soroka Medical Center - Internal Medicine Department, Beersheba
  - Edith Wolfson Medical Center | Internal Medicine Department, Holon
  - Hadassah University Medical Center (HUMC), Jerusalem
  - Health Corporation of Galilee Medical Center, Nahariya
  - Rabin Medical Center | Beilinson Hospital - Internal Medicine C Department, Petah Tikva
  - Health Corporation of the Ziv Medical Center (R.A.), Safed
- Italy (14):
  - Casa Sollievo della Sofferenza - Endocrinologia, San Giovanni Rotondo, Apulia
  - Azienda Ospedaliero Universitaria Parma - SC Nefrologia, Parma, Emilia-Romagna
  - ASL 4 Chiavarese, Chiavari, Liguria
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII - Malattie Endocrine e Diabetologia, Bergamo, Lombardy
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Endocrinologia, Milan, Lombardy
  - Ospedale San Raffaele s.r.l. - Medicina Generale Indirizzo Diabetologico ed Endocrino-Metabolico, Milan, Lombardy
  - Azienda Socio Sanitaria Territoriale Santi Paolo e Carlo_Ospedale S. Paolo - Gestione integrata della malattia Diabetica, Milan, Lombardy
  - Azienda Socio Sanitaria Territoriale Rhodense, Rho, Lombardy
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga - Malattie Metaboliche Diabetologia, Orbassano, Piedmont
  - Azienda Socio Sanitaria Locale N 2 Della Gallura - Diabetologia, Olbia, Sardinia
  - Azienda Ospedaliero Universitaria Pisana_Cisanello - Malattie Metaboliche e Diabetologia, Pisa, Tuscany
  - Azienda Ospedaliera Universitaria Integrata Verona_Borgo Roma - Endocrinologia, Diabetologia e Malattie del Metabolismo, Verona, Veneto
  - Università degli Studi "G. D'Annunzio" di Chieti - Endocrinologia, Chieti
  - Many Locations, Multiple Locations
- Japan (13):
  - Saiseikai Matsuyama Hospital, Matsuyama, Ehime
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Hirohata Naika Clinic, Kitakyushu, Fukuoka
  - Jiyugaoka Yamada Internal Medicine Clinic, Obihiro, Hokkaido
  - Naka Kinen Clinic, Naka, Ibaraki
  - Public Central Hospital of Matto Ishikawa | Clinical Trial Management Office, Hakusan, Ishikawa-ken
  - Fukui-ken Saiseikai Hospital, Fukui
  - Social Medical Corporation the Chiyukai foundation Fukuoka Wajiro Hospital, Fukuoka
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - Many Locations, Multiple Locations
  - Medical Corporation Taifukukai, Osaka Nishiumeda Clinic, Osaka
  - Osaka General Medical Center, Osaka
- Netherlands (4):
  - Meander Medisch Centrum, Amersfoort
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Gelre Ziekenhuizen, Apeldoorn
  - Albert Schweitzer Ziekenhuis | Dordwijk - Cardiology Department, Dordrecht
- South Korea (13):
  - Soon Chun Hyang University Cheonan Hospital, Cheonan, Chungcheongnam-do
  - Yonsei University Wonju Christian Hospital, Wŏnju, Gang''weondo
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggido
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - The Catholic University of Korea, Incheon St.Mary's Hospital, Incheon, Incheon Gwang''yeogsi
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Chung Nam National University Hospital, Daejeon
  - Korea University Ansan Hospital, Gyeonggi-do
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
- Spain (15):
  - Gerencia de Gestion Integrada A Coruna | Department of Endocrinology and Nutrition, A Coruña, A Coruña
  - Complejo Hospitalario Universitario de Ferrol | Hospital Naval - Unidad de Hipertensión Arterial, Ferrol, A Coruña
  - Hospital Principe de Asturias, Alcalá de Henares, Madrid
  - H. Costa del Sol (Marbella), Marbella, Malaga
  - Hospital Vithas Sevilla | Endocrinology Department, Castilleja de la Cuesta, Sevilla
  - Ciutat Sanitaria i Universitaria de la Vall d'Hebron, Barcelona
  - Hospital Quironsalud Barcelona | Internal Medicine Department, Barcelona
  - Hospital Universitario Virgen de las Nieves | Servicio de Endocrinologia y Nutricion, Granada
  - Hospital Clinico San Carlos, Madrid
  - Universidad Autonoma de Madrid (UAM) - Facultad de Medicina - Hospital Universitario Fundacion Jimenez Diaz (UAM-FJD), Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda | Clinical Pharmacology Department, Majadahonda
  - Hospital Universitario Virgen de la Victoria | Unidad de Investigacion Clinica - Endocrinology Department, Málaga
  - Many Locations, Multiple Locations
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia
- Taiwan (8):
  - Changhua Christian Hospital, Changhua
  - Chang Gung Memorial Hospital Kaohsiung, Kaohsiung City
  - Many Locations, Multiple Locations
  - Far Eastern Memorial Hospital | Nephrology Department, New Taipei City
  - Taipei Medical University - Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Agarwal R, Green JB, Heerspink HJL, McGill JB, Mottl A, Nangaku M, Rosenstock J, Rossing P, Vaduganathan M, Solis-Herrera C, Scott C, Li L, Brinker M, Aldworth C, Mann JFE. Risk of Hyperkalemia With Empagliflozin, Finerenone, or Both: Secondary Analysis of the CONFIDENCE Randomized Trial. J Am Coll Cardiol. 2025 Nov 7:S0735-1097(25)10035-1. doi: 10.1016/j.jacc.2025.10.049. Online ahead of print. PMID 41493296
- [Derived] Agarwal R, Green JB, Heerspink HJL, Mann JFE, McGill JB, Mottl A, Osonoi T, Pal A, Rossing P, Rosenstock J, Vaduganathan M, Li L, Li N, Scott C, Manjrekar P, Yamashita S, Nangaku M. Impact of Simultaneous Initiation of Finerenone and Empagliflozin on Urinary Albumin-to-Creatinine Ratio in Asia: Pre-Specified Analysis of CONFIDENCE. Clin J Am Soc Nephrol. 2026 Jan 1;21(1):72-82. doi: 10.2215/CJN.0000000865. Epub 2025 Sep 18. No abstract available. PMID 40965042
- [Derived] Vaduganathan M, Green JB, Heerspink HJL, Kim SG, Mann JFE, McGill JB, Mottl A, Nangaku M, Rosenstock J, Rossing P, Li L, Li N, Rohwedder K, Scott C, Agarwal R. Simultaneous initiation of finerenone and empagliflozin across the spectrum of kidney risk in the CONFIDENCE trial. Nephrol Dial Transplant. 2025 Dec 23;41(1):161-170. doi: 10.1093/ndt/gfaf160. PMID 40886054
- [Derived] Agarwal R, Green JB, Heerspink HJL, Mann JFE, McGill JB, Mottl AK, Rosenstock J, Rossing P, Vaduganathan M, Brinker M, Edfors R, Li N, Scheerer MF, Scott C, Nangaku M; CONFIDENCE Investigators. Finerenone with Empagliflozin in Chronic Kidney Disease and Type 2 Diabetes. N Engl J Med. 2025 Aug 7;393(6):533-543. doi: 10.1056/NEJMoa2410659. Epub 2025 Jun 5. PMID 40470996
- [Derived] Agarwal R, Green JB, Heerspink HJL, Mann JFE, McGill JB, Mottl AK, Rosenstock J, Rossing P, Vaduganathan M, Brinker M, Edfors R, Li N, Scheerer MF, Scott C, Nangaku M; CONFIDENCE investigators. COmbinatioN effect of FInerenone anD EmpaglifloziN in participants with chronic kidney disease and type 2 diabetes using a UACR Endpoint (CONFIDENCE) trial: baseline clinical characteristics. Nephrol Dial Transplant. 2025 Aug 1;40(8):1559-1569. doi: 10.1093/ndt/gfaf022. PMID 39916475
- [Derived] Rossing P. Experimental Designs for Multicomponent Interventions in Kidney and Cardiometabolic Diseases. J Am Soc Nephrol. 2024 Oct 1;35(10):1438-1441. doi: 10.1681/ASN.0000000000000449. Epub 2024 Jul 5. No abstract available. PMID 39078403
- [Derived] Zachariah T, Radhakrishnan J. Potential Role of Mineralocorticoid Receptor Antagonists in Nondiabetic Chronic Kidney Disease and Glomerular Disease. Clin J Am Soc Nephrol. 2024 Nov 1;19(11):1499-1512. doi: 10.2215/CJN.0000000000000540. Epub 2024 Jul 22. PMID 39037799
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — https://clinicaltrials.bayer.com/study/21839